CLINICAL TRIAL: NCT03563391
Title: A Prospective, Open Label, Multi-site Study in North America to Evaluate the Effects of a New Ready-to-feed, Nutrient Dense Formula on the Growth, Safety and Tolerance of Infants With Growth Failure
Brief Title: A Study to Evaluate the Effects of a New Formula on the Growth, Safety and Tolerance of Infants With Growth Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia North America (Industry)
Collaborators: Medical College of Wisconsin (Other); GI Care for Kids (Other); East Carolina University (Other); Wake Forest University Health Sciences (Other); Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CT17USCBUFG01
Record Dates: First submitted 2018-03-28; First posted 2018-06-20 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Growth Failure; Congenital Heart Disease
MeSH Terms: conditions — Failure to Thrive; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: A prospective, open-label, multi-site, growth, safety and tolerance study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of a new infant formula (Experimental): To evaluate the effects of a new formula on the growth, safety and tolerance of infants with growth failure
  Interventions: Other: New Infant Formula

INTERVENTIONS:
Other: New Infant Formula — New Infant Formula is a specialized, nutritionally complete, nutrient-dense infant formula specifically formulated for infants with growth failure.

SUMMARY:
This study is a prospective, open-label, multi-site, growth, safety and tolerance study to evaluate a NF (New Formula). A minimum of 45 evaluable infants with confirmed growth failure will be enrolled. Growth failure for 30 infants will be due to congenital heart disease and 15 infants due to other organic or non-organic causes. Study infants (in-patient or living with parents/ caregivers at home) will be fed the NF for a period of up through 16 weeks or until the time the infant subject meets criteria for switching to a lower calorie density formula, relative to baseline in infants with growth failure. Weight, height, head circumference and mid upper arm circumference will be measured regularly throughout the study. NF and other food intake, tolerance and stool diaries will be completed regularly. Serious adverse and adverse events will be monitored throughout the study. Infants will be evaluated, at each study visit, for criteria to switch to a lower calorie density formula. The primary objective is to improve weight-for-age z score relative to baseline. The secondary objectives are to improve weight-for-length, length-for-age, head circumference-for-age, mid upper arm circumference-for-age, weight velocity and length velocity z scores relative to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Infants must have attained term gestation (≥37 weeks of gestational age) at the time of screening
2. Infants, male or female, aged 1 through 8 months
3. Infants with congenital heart disease or other organic/non-organic cause of growth failure with a weight-for-length z score ≤ -1.0 or weight gain ≤ -2.0 z score based on WHO growth standards. (for weight gain metrics please see Appendix I): Weight gain (g) for boys and girls by age ( -2 z scores for weight velocity). Infants with Down syndrome must have a weight for length z-score ≤-1.0 z score. Infants with Down syndrome who meet the weight gain criterion (≤ -2.0 z-score weight gain) and have a weight for length z-score >-1.0 z-score will not be eligible for enrolment.
4. Infants expected to consume (or obtain via tube feeding), on average, 80% of their total energy intake from NF for 16 weeks
5. Infants from families who are willing and able to have anthropometrics taken at the required frequency as well as to comply with all other protocol requirements
6. Written informed consent from the parent/caregiver or legal guardian
7. Parent/caregiver or legal guardian must be able to read, write, and understand English

Exclusion Criteria:

1. Infants with known or suspected complex gastrointestinal anomalies or dysfunction, hepatic* or renal* dysfunction, or inherited metabolic disorders, congenital neurological insults, suspected or diagnosed conditions associated with malabsorption (e.g. cystic fibrosis)
2. Infants with known or suspected systemic or congenital infections (e.g. human immunodeficiency virus, HBV, HCV)
3. 3. Infants with known or suspected genetic conditions listed in Appendix VI and/or metabolic conditions known to interfere with growth or body dysmorphology that can interfere with obtaining standard anthropometric measurements (weight, length, head circumference, and mid upper arm circumference), with the exception of infants diagnosed with Down syndrome who may be enrolled in the study
4. Infants with known or suspected cow milk allergy or children who have received cow milk formula for 7 days or less
5. Infants expected to consume on average more than 20% of their energy intake from non-NF sources of nutrition: solids, expressed breast milk and /or parenteral nutrition.
6. Child feeding directly at the breast more than twice per day
7. Infants participating in any other studies involving investigational or marketed products concomitantly or within two weeks prior to the entry into the study. Infants participating in vaccination trials, who are only receiving follow-up blood monitoring, are not excluded.
8. Principal Investigator's uncertainty about the willingness or ability of the parent/caregiver or legal guardian to comply with the protocol requirements
9. Infants whose parent is younger than the legal age of consent
10. Infants born large for gestational age (LGA). LGA: Birth weight > 90th percentile for gestational age (please see chart in Appendix I)
11. Infants born small for gestational age (SGA). SGA: Birth weight < 10th percentile for gestational age (please see chart in Appendix I) * Note: For hepatic dysfunction, a conjugated bilirubin >2.0 mg/dL and for renal dysfunction child should not meet any of the pRIFLE criteria for renal disease (estimated creatinine clearance decreased by 25% by the Schwartz formula or urine output <0.5 mL/kg per hour over the previous 8 or more hours) or has chronic medical renal disease. In most children labs need not be obtained. These criteria only come into play when there is a consideration of liver or renal disease in the individual child.

Ages: 1 Month to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Change in weight-for-age z-score from baseline | 16 weeks
  weight for age z-score at 16 weeks (or at time of meeting criteria to switch to lower density formula if criteria is met prior to 16 weeks) and z-score at baseline

SECONDARY OUTCOMES:
Weight-for-length | 16 weeks
  z-score
Length-for-age | 16 weeks
  z-score
Head circumference-for-age | 16 weeks
  z-score
Mid upper arm circumference (MUAC)-for-age | 16 weeks
  z-score
Weight velocity | 16 weeks
  z-score
Length velocity | 16 weeks
  z-score

OTHER OUTCOMES:
Gastrointestinal tolerance | 16 weeks
  3-day diaries
Number of adverse events related to new infant formula (New Formula) | Up to 21 weeks starting from date of baseline visit
  Number of adverse events evaluated to be related to new infant formula (New Formula) using Adverse Events Decision Tree criteria

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Goday, MD, Principal Investigator — The Medical College of Wisconsin
Locations (5):
- United States (5):
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - GI Care for Kids, Atlanta, Georgia
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Medical College of Wisconsin, Milwaukee, Wisconsin